CLINICAL TRIAL: NCT06687993
Title: Acetylcholinesterase Inhibitor Treatment in Anorexia Nervosa: a Multicenter, Double-Blind, Placebo-Controlled Randomized Trial
Brief Title: Acetylcholinesterase Inhibitor in Anorexia Nervosa: Multicenter, Double-Blind, Placebo-Controlled Trial
Acronym: ANACh
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Université Paris Cité (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D22-P020; 2024-511681-37-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-30; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-07

CONDITIONS: Anorexia Nervosa Restricting Type
Keywords: anorexia nervosa; eating disorders; donepezil; habits
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders; Habits | interventions — Donepezil

STUDY DESIGN:
Intervention Model Description: Multicenter, superiority study, in double-blind, randomized, parallel groups, controlled versus placebo, in using a sequential adaptive design by band.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind design. Comparative analyzes will be carried out blindly
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- donepezil 2.5 mg (Experimental): donepezil 2.5 mg daily for 90 days
  Interventions: Drug: Donepezil 2.5 mg
- donepezil 5 mg (Experimental): donepezil 5 mg daily for 90 days
  Interventions: Drug: Donepezil 5 mg
- placebo (Placebo Comparator): placebo daily for 90 days
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Donepezil 2.5 mg — 2.5 mg daily oral intake for 90 days
  Other Names: Donepezil chlorhydrate
  Arms: donepezil 2.5 mg
Drug: Donepezil 5 mg — 5 mg daily oral intake for 90 days
  Other Names: Donepezil chlorhydrate
  Arms: donepezil 5 mg
Drug: Placebo Comparator — daily oral intake for 90 days
  Other Names: Placebo
  Arms: placebo

SUMMARY:
The goal of this clinical trial is to learn if the daily take of donepezil can treat adult patient suffering from anorexia nervosa. The main question it aims to answer is : do daily donepezil intake permit weight gain and reduction of food restriction rituals ? The treatment is a capsule comprising a drug limiting the degradation of a neurotransmitter called acetylcholine. This treatment has long been used to treat certain cognitive disorders. Researchers will compare two drug dosage and a look-alike capsule that contains no drug to see if the dose has an impact on the effect. Participants will take one capsule per day for three months will have regular hospital visits for cognitive and metabolic tests.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Presence of the 3 DSM-V criteria for Anorexia Nervosa
* Restrictive subtype of Anorexia Nervosa according to DSM-5
* Body Mass Index between 15 and 18.5 kg/m²
* Aged 18 to 65 years
* Resting heart rate > or = 40 bpm
* Use of a highly effective contraceptive method
* Affiliation or entitlement to a Health Insurance scheme
* Prior free, informed, and written consent

Exclusion Criteria:

* Presence of one or more somatic criteria for hospitalization according to french HAS 2010 guidelines
* Past diagnosis of anorexia nervosa with binge-eating/purging type
* Past diagnosis of bulimia nervosa
* Past diagnosis of binge-eating disorder
* Associated diagnosis of schizophrenia and/or persistent delusional disorder and/or bipolar disorder
* History of asthma or obstructive bronchopulmonary disease
* History of peptic ulcer disease or concurrent treatment with non-steroidal anti-inflammatory drugs
* History of epileptic disorders
* Renal insufficiency (glomerular filtration rate less than 60 mL/min according to the MDRD formula)
* Hepatic insufficiency or transaminase levels greater than 5 times the normal upper limit
* Conductance disorder characterized by electrocardiogram
* QTc according to Bazett's formula greater than 480 ms on electrocardiogram
* Current or recent (within three weeks prior to inclusion) psychotropic treatment (including antidepressants, to avoid interaction/potentiation in this population)
* Treatment involving the following cytochromes: P450, P3A4, P2D6
* Known hypersensitivity to donepezil hydrochloride, piperidine derivatives, or any excipients of the investigational drug
* Pregnant or breastfeeding woman
* Person under legal protection measures
* Person under guardianship measures

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2030-02 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Effect on Body Mass Index in adult women suffering from anorexia nervosa | Before (D0) and after 90 days of treatment
  Difference of Body Masse Index between inclusion (D0) and the end of treatment (D90)

SECONDARY OUTCOMES:
Effect on eating disorder symptomatology in adult women suffering from anorexia nervosa: difference of Eating Disorder Examination Questionnaire (EDE-Q) score | Before (D0) and after 90 days of treatment
  The Eating Disorder Examination Questionnaire (EDE-Q) is a self-report measure used to assess the severity of eating disorder symptoms. The scale consists of four subscales: Restraint, Eating Concern, Shape Concern, and Weight Concern, along with a Global score.
  Scale Range: Each subscale score and the Global score range from 0 to 6. Score Interpretation: Higher scores indicate greater severity of eating disorder symptoms. A higher score reflects a worse outcome in terms of eating disorder symptom severity.
Effects on habits learning in adult women suffering from anorexia nervosa: difference of phase 3 of slips-of-action neurocognitive test | Before (D0) and after 90 days of treatment
  The Slips-of-Action Neurocognitive Test is a measure designed to assess cognitive control, focusing on the ability to inhibit responses that are no longer contextually appropriate. In Phase 3 of this test, participants must withhold previously learned responses as the rules change, evaluating their inhibitory control capacity.
  Scale Range: Scores in Phase 3 range from 0 to 20, representing the number of errors (or "slips") made during the test.
  Score Interpretation: Higher scores reflect a greater number of inhibitory errors, indicating reduced cognitive control. Thus, a higher score represents a worse outcome in terms of inhibitory control performance.
Effect on balance between goal-directed behaviors and habits in adult women suffering from anorexia nervosa: difference of total score in Self-Report Habit Index | Before (D0) and after 90 days of treatment
  The Self-Report Habit Index (SRHI) is a tool used to measure the strength of habitual behaviors. It assesses habits across various domains, providing a total score that reflects the extent to which a behavior has become automatic.
  Scale Range: The total score ranges from 0 to 42, with higher scores indicating stronger habitual behavior.
  Score Interpretation: A higher score suggests a more entrenched habit, reflecting a stronger habitual response. Thus, higher scores indicate a worse outcome if the goal is to reduce the habitual behavior.
Effect on cognitive flexibility in adult women suffering from anorexia nervosa: difference in Wisconsin Card Sorting Test | Before (D0) and after 90 days of treatment
  The Wisconsin Card Sorting Test (WCST) assesses cognitive flexibility and executive function by measuring an individual's ability to adapt to changing rules and shift cognitive strategies.
  Scale Range: Scores are typically reported as the number of perseverative errors, ranging from 0 to a maximum depending on the number of trials (typically 128).
  Score Interpretation: Higher scores indicate more errors and reflect poorer cognitive flexibility. Therefore, a higher score represents a worse outcome in terms of executive functioning.
Effect on cognitive flexibility in adult women suffering from anorexia nervosa: difference in Trail Making Test B-A, Brixton Test | Before (D0) and after 90 days of treatment
  The Trail Making Test (TMT) is used to assess cognitive processing speed, flexibility, and task-switching abilities. TMT B-A represents the difference in time taken to complete Part B (which involves both numbers and letters) compared to Part A (numbers only).
  Scale Range: The B-A score is expressed in seconds, typically ranging from 0 to several hundred seconds depending on the individual's performance.
  Score Interpretation: Higher scores indicate slower processing and greater difficulty with task switching, representing a worse outcome for cognitive flexibility and processing speed.
Effect on compulsive and obsessive in adult women suffering from anorexia nervosa: difference in Yale-Brown Obsessive Compulsive Scale | Before (D0) and after 90 days of treatment
  The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is a clinician-administered tool used to assess the severity of obsessive-compulsive symptoms, measuring both obsessions and compulsions.
  Scale Range: The total score ranges from 0 to 40, with subscales for obsessions and compulsions each ranging from 0 to 20.
  Score Interpretation: Higher scores indicate greater severity of OCD symptoms. Thus, a higher total score reflects a worse outcome in terms of obsessive-compulsive symptom severity.
Effect on main eating disorder dimensions in adult suffering from anorexia nervosa: difference in subdimensions on EDE-Q and Eating Disorder Iventory 3 | Before (D0) after 90 days of treatment and 90 days after stopping treatment
  Eating Disorder Inventory-3 (EDI-3) Subdimensions The EDI-3 measures psychological traits associated with eating disorders through 12 subscales, including Drive for Thinness, Bulimia, Body Dissatisfaction, Low Self-Esteem, Personal Alienation, Interpersonal Insecurity, Interpersonal Alienation, Interoceptive Deficits, Emotional Dysregulation, Perfectionism, Asceticism, and Maturity Fears.
  Scale Range: Each subscale has a score range of 0 to 16, though the maximum score can vary slightly depending on the specific items within each subscale.
  Score Interpretation: Higher scores indicate greater severity of the particular trait or symptom associated with eating disorders. Therefore, higher scores across subscales reflect a worse outcome regarding eating disorder psychopathology.
Effect on depressive and anxious symptoms in adult women suffering from anorexia nervosa: difference on Hospital Anxiety and Depression Scale (HADS) | Before (D0) and after 90 days of treatment
  The Hospital Anxiety and Depression Scale (HADS) is a self-report measure designed to assess levels of anxiety and depression in patients, particularly in hospital settings. The scale consists of two subscales: Anxiety (HADS-A) and Depression (HADS-D).
  Scale Range: Each subscale (HADS-A and HADS-D) has a score range from 0 to 21, with the total score ranging from 0 to 42.
  Score Interpretation: Higher scores indicate more severe symptoms of anxiety or depression. Thus, higher scores on each subscale, or the total score, represent worse outcomes in terms of anxiety and depression severity.
Measure the toxicity and tolerance of donepezil in adult women suffering from anorexia nervosa | D3, D5, D30, D90
  Difference of frequency of adverse effects
Biological factors associated with response to treatment | Before (D0) and after 90 days of treatment
  Gut microbiome diversity (Simpson, Shannon and Chao1) and nutritional plasmatic biomarkers

IPD SHARING:
Plan to Share IPD: Undecided